CLINICAL TRIAL: NCT00094185
Title: Clotting Genetic Variants, Hormones, and Venous Thrombosis
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1277; R01HL073410-01 (NIH)
Record Dates: First submitted 2004-10-15; First posted 2004-10-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Cardiovascular Diseases; Thromboembolism
MeSH Terms: conditions — Cardiovascular Diseases; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- General: No intervention

SUMMARY:
To identify genetic variants in 12 key blood clotting proteins that may modify the risk of venous thromboembolism in users of hormone replacement therapy.

DETAILED DESCRIPTION:
BACKGROUND:

Venous thromboembolism (VTE) occurs commonly in adults and risk increases 3-fold among users of hormone replacement therapy (HRT), oral contraceptives (OC), and selective estrogen receptor modulators (SERMs). Epidemiologic data suggest that genetic variation in the pro-coagulant, anti-coagulant, and fibrinolytic pathways may modify the risk of VTE in women, especially in the presence of hormone use. The primary aim of this study is to identify genetic variants in 12 key clotting proteins that may modify the risk of VTE independently, through gene-gene interactions, and in the presence of HRT, OC, or SERM use. Proteins include thrombomodulin, protein C, endothelial protein C receptor, protein S, antithrombin III, tissue activatable fibrinolysis inhibitor (TAFI), tissue plasminogen activator (TPA), and factors VIII, IX, X, and XlII A and B. Secondary aims are to determine if levels of TAFI antigen, TPA antigen, activated protein C resistance, and D-dimer serve as intermediate phenotypes for gene-drug interactions and VTE risk. The setting for this study is Group Health Cooperative (GHC) of Puget Sound, a health maintenance organization in the Pacific Northwest. This study is part of an on going, case-control study addressing the effects of genetic variants on drug safety, particularly cardiovascular endpoints.

DESIGN NARRATIVE:

The primary aim of this case-control study is to identify genetic variants in 12 key blood clotting proteins that may modify the risk of venous thromboembolism independently, through gene-gene interactions, and in the presence of hormone replacement therapy, oral contraceptives, or selective estrogen receptor modulators use. Proteins include thrombomodulin, protein C, endothelial protein C receptor, protein S, antithrombin III, tissue activatable fibrinolysis inhibitor (TAFI), tissue plasminogen activator (TPA), and factors VIII, IX, X, and XlII A and B. Secondary aims of the study are to determine if levels of TAFI antigen, TPA antigen, activated protein C resistance, and D-dimer serve as intermediate phenotypes for gene-drug interactions and VTE risk. The setting for this study is the Group Health Cooperative (GHC) of Puget Sound, a health maintenance organization in the Pacific Northwest. This study is part of an on going, case-control study addressing the effects of genetic variants on drug safety, particularly cardiovascular endpoints.

All inpatient and outpatient VTE events occurring between 1/1/1995 and 12/31/2007 among women 18 to 89 years of age will be eligible for this study. Controls will be a random selection of women from GHC matched on age, hypertension status, and calendar year. Medical records will be reviewed to determine study eligibility and to collect V'i'E risk factor information. Hormone and SERM use will be ascertained from the GHC pharmacy database. Phlebotomy will be performed on surviving cases and controls to collect plasma samples and genetic information. Logistic regression analyses will determine which haplotypes of key elements in the clotting pathways modify the association between hormones or SERMSs and VTE risk. The identification of common genetic variants that either increase or decrease VTE risk independently or in the presence of hormone or SERMs will help to inform clinicians and their female patients about the personal safety of hormone use.

The Seattle Program for Genomics Applications (PGA) will identify single nucleotide polymorphisms (SNPs) in the 12 candidate genes and use linkage disequilibrium to generate haplotypes. A group at the Leiden University Medical Center will perform the genotyping of the study population.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2004-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Venous Thrombosis | Retrospective
  Incidence of venous thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Smith, Study Chair — University of Washington